CLINICAL TRIAL: NCT04229342
Title: Comparison of Gastroesophageal Reflux Between Conventional Versus Oblique Fibers Sparing Endoscopic Myotomy for Achalasia Cardia - A Randomized Controlled Trial
Brief Title: Post-POEM GERD in Patients Undergoing Conventional Versus Oblique Fibers Sparing Posterior Myotomy for Achalasia Cardia
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Principal Investigator, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POEM001
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2020-10

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): In the "conventional group", standard posterior myotomy will be performed and the sling or the oblique fibers will not be spared beyond the gastroesophageal junction.
  Interventions: Procedure: Per-oral endoscopic myotomy
- Oblique or sling fiber sparing group (Experimental): In the oblique or sling fiber group, only the circular muscle fibers will be severed selectively and the sling fibers will be spared
  Interventions: Procedure: Per-oral endoscopic myotomy

INTERVENTIONS:
Procedure: Per-oral endoscopic myotomy — Per-oral endoscopic myotomy (POEM) is an endoscopic modality for the management of achalasia cardia. In this study, we will evaluate the impact of two different techniques of posterior POEM on the incidence of gastroesophageal reflux disease (GERD).
  Posterior POEM will be performed using the standard technique. The myotomy beyond the GEJ will be different in the two groups. In one group, the sling fibers will not be spared from dissection and in the second group, the sling fibers will be selectively spared from myotomy.

SUMMARY:
In this study, we will evaluate the incidence of reflux esophagitis between two different techniques of posterior per-oral endoscopic myotomy (POEM) i.e. conventional POEM versus oblique/ sling fiber sparing POEM. This is a randomized trial where the patients with idiopathic achalasia will be randomized in two groups in 1:1 fashion into groups.

DETAILED DESCRIPTION:
In this randomized trial, patients with idiopathic achalasia will undergo POEM using two techniques as follows. In the first technique, a conventional posterior POEM will be performed where the sling or oblique fibers will not be spared during POEM. Sling or oblique fibers will be recognized using the configuration of fibers below the gastroesophaeal junction and by identifying the border between the sling fibers and the circular fibers which is formed by the penetrating vessels. In the second group (Oblique fiber group), the sling fibers will be selectively spared and only the circular fibers will be spared.

The other steps of the POEM procedure will be the same as described in the standard technique of POEM. These include submucosal injection of saline mixed with indigo carmine dye, mucosal incision, submucosal tunneling using triangular knife in spray coagulation mode (Effect 2, Watts 50), myotomy extending upto 2-4 cm below the gastroesophageal junction and the closure of mucosal incision using endoclips.

Post POEM management: All the patients will be kept nil per oral for about 24-hours after the procedure. A timed barium swallow will be performed the next day and oral liquids will be started. A soft puried diet will be started from day 3 onwards.

Oral proton pump inhibitors (PPIs) equivalent to 40 mg of Pantoprazole per day will be prescribed to all the patients unless a contraindication exists.

Follow-up: The first evaluation will be performed at 2-months after POEM. During this evaluation, the following parameters will be recorded: symptom relief, reflux symptoms, and esophageal acid exposure. PPIs will be stopped for 1-2 weeks prior to the evaluation of GERD.

Subsequent evaluation will be at 6-months for reflux symptoms and symptoms of achalasia using Eckardt scores.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 1 and 2 achalasia with Eckardt score >3 (0-12 scale achalasia).
2. Patients with age 18-75 years.
3. Patients who are treatment naïve or have a history of pneumatic balloon dilatation.
4. Patients who are willing and able to comply with the study procedures and provide written informed consent form to participate in the study

Exclusion Criteria:

1. Patients with type 3 achalasia cardia or any other esophageal motility disorder,
2. Patients who have undergone previous surgery of the esophagus or stomach,
3. Patients with active severe esophagitis,
4. Patients with large lower esophageal diverticula,
5. Patients with large ( > 3cm ) hiatal hernia,
6. Patients with sigmoid oesophagus,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Significant Reflux Esophagitis, Los Angeles grade (≥grade B) | 8 weeks
  Assessment of reflux esophagitis will be done at 8 weeks post procedure using Los Angeles grading system (grade A to D)

SECONDARY OUTCOMES:
Clinical Success, Eckardt Score (minimum: 0, maximum: 12), Eckardt Score≤3: success, >3: failure | 8 weeks
  Clinical success will be evaluated using Eckardt scores
Clinical success using Eckardt Score (minimum:0, maximum: 12) | 6 months
  Clinical success will be evaluated using Eckardt scores. Eckardt Score≤3 will be considered as clinical success and >3 will be considered as clinical failure
Esophageal manometry | 8 weeks
  Esophageal manometry will be performed at 8 weeks and Integrated relaxation pressure will be calculated and presented in mmHg 5. Change in IRP pressure by Manometry ( Assessed at pre procedure & 8 weeks).
Barium column height on Timed barium swallow; Success: >50% reduction in barium column height | 2 months
  Timed barium swallow will be performed after POEM procedure and Esophageal emptying will be seen and compared with pre-POEM timed barium esophagogram
Esophageal acid exposure, Acid exposure time>6 abnormal, <4: normal, 4-6: inconclusive | 8 weeks
  24-hour pH impedance study will be performed at 8-weeks and esophageal acid exposure will be calculated
Reflux Symptoms, GERD HRQL score (minimum score: 0, maximum score: 50) | 8-weeks
  The symptoms of gastroesophageal reflux will be evaluated using symptom scores.
Gastroesophageal reflux with DeMeester score at 8-weeks: DeMeester score≥14.7 abnormal, <14.7: normal | 8 weeks
  DeMeester scores will be calculated at 8 weeks after the POEM procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Vincy Chandran, MBBS,MD, Principal Investigator — Asian Institute of Gastroenterology Hospital
Locations (1):
- Asian institute of Gastroenterology/AIG Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nabi Z, Chandran V, Basha J, Ramchandani M, Inavolu P, Kalpala R, Goud R, Jagtap N, Darisetty S, Gupta R, Tandan M, Lakhtakia S, Kotla R, Devarasetty R, Rao GV, Reddy DN. Conventional versus oblique fiber-sparing endoscopic myotomy for achalasia cardia: a randomized controlled trial (with videos). Gastrointest Endosc. 2024 Jan;99(1):1-9. doi: 10.1016/j.gie.2023.08.007. Epub 2023 Aug 19. PMID 37598863